CLINICAL TRIAL: NCT01568528
Title: Oxytocin as Adjunctive Treatment of Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Atlanta VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Erica Duncan, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00052127
Record Dates: First submitted 2012-03-28; First posted 2012-04-02 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Oxytocin (Experimental): The intranasal oxytocin intervention will be the administration of OT intranasally at a dose of three 4 IU puffs per nostril for a total dose of 24 IU. Each puff is 0.1ml in volume so the total volume administered will be 0.6 ml intranasally. This dose has been used in a number of other similarly designed challenge studies examining the effects of a single dose of OT (Kirsch et al. 2005; Kosfeld et al. 2005; Guastella et al. 2008a; Guastella et al. 2008b; Rimmele et al. 2009; Andari et al. 2010).
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Intranasal placebo The PBO/control will consist of the OT vehicle administered as three puffs in each nostril. Each puff is is 0.1ml in volume so the total volume administered will be 0.6 ml intranasally.
  Treatment assignment will be by random allocation in blocks of six. Both experimenters and subjects will be blind to the treatment they are receiving.
  Interventions: Drug: Placebo
- Healthy Controls (Other): Participants who have no psychiatric diagnosis and will be controls for this project. These controls will not receive oxytocin or placebo. They will only receive psychiatric screening interview, MATRICS Consensus Cognitive Battery (MCCB) assessment, urine drug screen, vision testing, and the three social cognition tasks.
  Interventions: Other: Control

INTERVENTIONS:
Drug: Oxytocin — OT intervention will be administration of OT intranasally at a dose of three 4 IU puffs per nostril for a total dose of 24 IU. This dose has been used in a number of other similarly designed challenge studies examining the effects of a single dose of OT (Kirsch et al. 2005; Kosfeld et al. 2005; Guastella et al. 2008a; Guastella et al. 2008b; Rimmele et al. 2009; Andari et al. 2010).
  Other Names: Syntocinon
  Arms: Oxytocin
Drug: Placebo — The PBO/control will consist of the OT vehicle only delivered as 3 puffs of saline per nostril for a total of 6 puffs. Each puff contains 0.1 ml in volume, so the total delivered will be 0.6 ml intranasally.
  Other Names: Inactive vehicle
  Arms: Placebo
Other: Control — Participants who have no psychiatric diagnosis and will be controls for this project. These controls will NOT receive oxytocin or PBO. They will only receive psychiatric screening interview, MCCB Consensus Cogntive Battery assessment, urine drug screen, vision testing, and the three social cognition tasks.
  Arms: Healthy Controls

SUMMARY:
The focus of the current project is to advance our understanding of the effects of oxytocin (OT) on components of social cognition in schizophrenia (SCZ). Despite the rapid increase in our understanding of the role of OT in rodent models of social behavior and an explosion of interest in the prosocial effects of OT in healthy controls, little work has been done to dissect the potential effects of OT on SCZ subjects with social deficits. Social deficits are a crucial aspect of the functional impairments that limit the rehabilitation of patients with SCZ. In particular, SCZ patients with enduring negative symptoms (deficit syndrome, Kirkpatrick et al. 1989) have prominent social deficits as a core feature of this subtype of the illness. Our currently available medications do very little to improve these social deficits. Hence it is of utmost public health importance to address the knowledge gap regarding the potential of OT to improve social function in this illness. Intact social function depends on the competent functioning of several cognitive domains that subserve perception of social cues and the generation of motivated social behavior. We propose to conduct a pharmacological challenge study of OT vs. placebo administration to study the effects of OT on specific components of social cognition in male deficit syndrome SCZ subjects.

Primary Hypothesis: Intranasal OT will improve social cognition in subjects with deficit syndrome SCZ.

DETAILED DESCRIPTION:
Specific Aim 1: Administer OT intranasally vs. placebo in a parallel group double-blind design to 40 deficit syndrome SCZ subjects. Following OT or placebo (PBO) dosing, components of social cognition will be assessed as follows.

1. Evaluate the salience of social cues by the measurement of visual scan paths during gaze at pictures of faces.
2. Evaluate sensitivity to social reward by means of a computerized social reward ball-tossing task that assays social interactions in response to social reward.
3. Evaluate social cognition by means of testing the ability to correctly identify emotion from pictures of faces (Facial Emotion Identification Test, FEIT).

BACKGROUND

Impaired social functioning is an important symptom in SCZ SCZ is a chronic severe psychotic illness that affects two to three million Americans, over 100,000 of whom are veterans (Owen et al. 2004). There are several key symptom domains that characterize the illness. Positive symptoms (such as hallucinations and delusions) are at least somewhat responsive to antipsychotic medication in a majority of patients. Negative symptoms such as poor motivation, anhedonia, poor social function, and poor occupational function are poorly responsive to medication or other currently available treatments. The deficit syndrome has been defined as a complex of these negative symptoms that endure throughout the course of a schizophrenia patient's disease (Kirkpatrick et al. 1989). The social impairments seen in these patients are core deficits that have been linked to poor functional outcomes (Couture et al. 2006; Fett et al. 2011). Furthermore, deficits in social cognition have been proposed to underlie and contribute significantly to impaired social functioning (Kern et al. 2008; Green et al. 2008). An underlying hypothesis of this work is that if social cognition could be effectively treated, these patients would improve their social and functional outcomes, potentially enabling them to achieve occupational competence, sustain stable independent living, and lead more fulfilling independent lives. Thus our understanding and treatment of the social impairments of SCZ is very important from a public health perspective.

OT effects on social cognition and behavior Studies in rodents demonstrate a critical role for the neuropeptide OT in social bonding (Young et al. 2005). A large and rapidly growing translational literature indicates that this neuropeptide may also play a prosocial role in human behavior. The prosocial effects of OT administration have already been extensively reviewed in the literature (Striepens N et al., 2011). In the area of trust and altruism, studies utilizing a variety of economic and cooperation paradigms indicate that OT enhances trusting and social cooperation (Baumgartner T et al., 2008; De Dreu CK et al., 2010; Declerck CH et al., 2010; Kosfeld M et al., 2005; Mikolajczak M et al., 2010; Zak PJ et al., 2007). Feelings of empathy to others were enhanced with OT in three studies (Domes et al. 2007; Bartz et al. 2010; Hurlemann et al. 2010). Several studies indicate that OT increases the ability of healthy controls to identify emotion in faces (Di Simplicio et al. 2009; Fischer-Shofty et al. 2010, Marsh et al. 2010). There are reports using memory paradigms, in which OT administration induced enhanced recall of faces after OT (Savaskan et al. 2008; Rimmele et al. 2009), although an earlier study found no improvement (Ferrier et al. 1980). OT administration also increased recall of social words (Unkelbach et al. 2008). There is some indication that OT effects on recall are specific to emotional stimuli since several studies in healthy controls found that OT did not improve memory for nonsocial stimuli (Bruins J et al., 1992; Fehm-Wolfsdorf G et al., 1984; Geenen V et al., 1988; Kennett DJ et al., 1982).

OT as potential treatment in SCZ Several lines of reasoning suggest that OT could be helpful as adjunct treatment of SCZ.

1. Patients with SCZ have altered OT levels compared to healthy controls (Linkowski et al. 1984; Beckmann et al. 1985; Legros et al. 1992; Goldman et al. 2008; Keri et al. 2009).
2. fMRI in concert with intranasal OT administration was associated with reduced blood-oxygen-level-dependent (BOLD) activation in the amygdala during presentation of fearful/threatening faces and scenes (Kirsch et al. 2005). This study gives indirect support to the idea that OT may ameliorate paranoia in patients with SCZ.
3. The negative symptoms of SCZ include social isolation, autism, and amotivation for social engagement. There is face validity to the notion that OT could help with these symptoms in virtue of its pro-social action.
4. To date there are three published placebo controlled trials of OT in SCZ. In the first study, OT was given in a placebo-controlled double-blind randomized crossover design (Feifel et al. 2010). In this study of fifteen completers, the Positive and Negative Symptom Scale (PANSS) and the Clinical Global Impressions scale (CGI) were used as outcome measures. OT added to antipsychotic treatment resulted in a significant improvement in positive symptoms, as measured by the PANSS total score, PANSS positive symptom subscale, PANSS negative symptom subscale, and the CGI. The effect size for these changes ranged from 0.40 for PANSS positive symptoms to 0.74 for the CGI. Furthermore, treatment with OT was well tolerated, with no significant differences between OT and placebo in rates of adverse effects nor in blood chemistry (Feifel et al. 2010). This same group published a second paper indicating an improvement in verbal memory in SCZ subjects following three weeks of twice daily OT (Feifel et al. 2012). The third study reports that two weeks of OT reduced psychotic symptoms and improved performance in a Theory of Mind task (Pedersen et al. 2011).

Dissecting components of social impairment in SCZ Intact social competence depends on adequate function in several cognitive domains that subserve perception of social cues and motivated social behavior. We propose to interrogate these composite domains after administration of OT vs. placebo in this project.

i. Eye tracking. Relevant social cues must be of sufficient salience to command attention. This aspect of social cognition has been investigated by means of visual scan path paradigms that quantify the amount of time a subjects spends looking at the eyes and mouth regions of pictures of faces presented while the position of the eyes is tracked. The amount of eye gaze is predictive of a subject's ability to correctly identify emotions and meaning in others (Haxby et al. 2002). A single dose of OT significantly increases the amount of eye gaze in healthy controls (Guastella et al. 2008a) and in high functioning subjects with autism spectrum disorders (Andari et al. 2010). SCZ subjects have abnormalities in visual scan paths while viewing pictures of faces (Phillips and David 1997; Loughland et al. 2002a). Thus we hypothesize that OT will increase gaze at the eyes in subjects with deficit syndrome SCZ (Specific Aim 2a).

ii. Social Reward Ball-Tossing Task. Social stimuli must be sufficiently rewarding to motivate decision-making and behavior. This aspect of social function has been investigated with a computerized social interaction game that assays the effects of social reinforcement on decision-making. In a task developed by Andari et al. (2010) that was derived from an earlier task by Williams et al. (2000), subjects engage in a computerized version of a ball-toss game in which three fictional partners vary the proportion of times they throw the ball back to the subject. The outcome measure of interest was the choices made by the subject regarding to which fictional player they would throw the ball. In a study of high functioning autism spectrum subjects, OT administration selectively enhanced return of the ball to the most socially cooperative fictional partner (Andari et al. 2010). This result was interpreted as evidence that OT enhances appropriate behavioral responses to the social reward of reciprocity. We hypothesize that OT administration will enhance socially reinforced behavior in subjects with deficit syndrome SCZ (Specific Aim 2b).

iii. Facial Emotion Identification Task (FEIT). The socially competent person must be able to correctly identify the emotions in others in order to respond appropriately during social communication. The correct identification of emotions in others is a key aspect of social cognition that has been linked to functional outcomes in SCZ (Couture et al. 2006). This aspect of social cognition has been investigated in paradigms that query the subjects on identifying emotions displayed in pictures. Most studies in the literature report that patients with SCZ are deficient in the correct identification of emotions displayed in pictures of faces (Addington et al. 2006; Bigelow et al. 2006; van't Wout et al. 2007; Averbeck et al. 2012 and see review in Couture et al. 2006), although not all studies have found such impairments (de Achaval et al. 2010). The classic series of pictures of faces introduced by Eckman and Friesen (1976) have been used in many studies of affect recognition, but other series of pictures have also been utilized (Erwin et al. 1992; Kerr and Neale 1993). OT administration has been shown in two studies to increase the correct identification of emotions in faces in subjects with SCZ (Goldman et al. 2011; Averbeck et al. 2012). We hypothesize that deficit syndrome SCZ subjects will exhibit improvement in facial emotion recognition after administration of OT (Specific Aim 2c).

ELIGIBILITY:
Subjects for the study will be forty male VA patients with a diagnosis of schizophrenia. Diagnosis will be determined using the Structured Clinical Interview for DSM-IV Axis I Disorders/SCID-P (Spitzer et al. 1992). Subjects must be categorized as having a primary deficit syndrome on the Kirkpatrick Schedule for the Deficit Syndrome (Kirkpatrick et al. 1989).

Additional inclusion criteria:

1. Subjects must be between 18 and 65 years old at the time of study screening.
2. Subjects must demonstrate adequate decisional capacity, in the judgment of the consenting study staff member, to make a choice about participating in this research study.
3. Subjects must have been psychiatrically and medically stable for 8 weeks prior to consent in the judgment of the Principal Investigator.
4. Subjects must have been maintained on a stable treatment of antipsychotics and/or other concomitant psychotropic treatment for at least 6 weeks prior to consent.
5. Subjects must have no more than a moderate severity rating on hallucinations and unusual thought content as shown by a score of ≤ 4 on the Positive and Negative Symptoms Scale (PANSS).
6. Subjects must be able to validly complete the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery (MCCB), in the judgment of the consenting study staff person.
7. Subjects must have the visual, auditory, and motor capacity to use the computer software in the judgment of the consenting study staff person. Visual acuity must be at least 20/30 corrected.
8. Subjects must have a minimal level of extrapyramidal symptoms as shown by a Simpson-Angus Scale total score of no more than 6.
9. Subjects must have a minimal level of depressive symptoms as shown by a Calgary Depression Scale (CDSS) total score of no more than 10.

Exclusion criteria:

1. Female sex
2. History of bipolar disorder
3. Active substance dependence within the prior 30 days (cigarette smoking is allowed)
4. Has had a psychiatric hospitalization in the 8 weeks prior to consent.
5. Suicidal or homicidal ideation in the previous six months
6. Subjects who have answered 'yes' to Question 5 (Active Suicidal Ideation with Specific Plan and Intent) on the Columbia-Suicide Severity Rating Scale, C-SSRS, or who have answered 'yes' to any of the suicide-related behaviors (actual attempt, interrupted attempt, aborted attempt, preparatory act or behavior) on the C-SSRS "Suicidal Behavior" portion shall be excluded from the study if ideation or behavior occurred within one month of consent. Subjects excluded for this reason will be referred for appropriate treatment.
7. History of mental retardation or pervasive developmental disorder
8. History of neurological disorder (e.g., traumatic brain injury, seizure disorder, Parkinson's Disease, dementia), loss of consciousness for more than 10 minutes due to head trauma, known HIV infection, or AIDS
9. Treatment with a benzodiazepine in the two weeks prior to consent.

Control Participants:

Inclusion Criteria:

* Male
* Ages 18-65

Exclusion Criteria:

* Female
* History of a psychotic disorder, or depression requiring medication
* Active substance abuse or dependence within the prior 30 days
* Medical admission within the past six months

Criteria to rule out subjects with medical problems likely to present a confound:

* Known HIV infection or AIDS
* History of TBI
* Seizure disorder
* Known Alzheimer's Disease or other dementia
* Minimal cognitive impairment (MCI)
* Parkinson's Disease
* Unstable medical condition

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-03; Primary Completion 2017-03-15 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica J Duncan, MD, Principal Investigator — Emory University
Locations (1):
- Atlanta VA Medical Center, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young LJ, Murphy Young AZ, Hammock EA. Anatomy and neurochemistry of the pair bond. J Comp Neurol. 2005 Dec 5;493(1):51-7. doi: 10.1002/cne.20771. PMID 16255009
- [Background] Andari E, Duhamel JR, Zalla T, Herbrecht E, Leboyer M, Sirigu A. Promoting social behavior with oxytocin in high-functioning autism spectrum disorders. Proc Natl Acad Sci U S A. 2010 Mar 2;107(9):4389-94. doi: 10.1073/pnas.0910249107. Epub 2010 Feb 16. PMID 20160081
- [Background] Guastella AJ, Mitchell PB, Dadds MR. Oxytocin increases gaze to the eye region of human faces. Biol Psychiatry. 2008 Jan 1;63(1):3-5. doi: 10.1016/j.biopsych.2007.06.026. Epub 2007 Sep 21. PMID 17888410
- [Background] Mueser KT, Doonan R, Penn DL, Blanchard JJ, Bellack AS, Nishith P, DeLeon J. Emotion recognition and social competence in chronic schizophrenia. J Abnorm Psychol. 1996 May;105(2):271-5. doi: 10.1037//0021-843x.105.2.271. PMID 8723008
- [Derived] Andari E, Massa NM, Fargotstein MD, Taylor NB, Halverson DM, Owens AV, Currin DL, Bhattacharya A, Gitman D, Cuthbert BC, Young LJ, Duncan EJ. Effects of Oxytocin on Emotion Recognition in Schizophrenia: A Randomized Double-Blind Pilot Study. J Clin Psychopharmacol. 2021 Mar-Apr 01;41(2):103-113. doi: 10.1097/JCP.0000000000001367. PMID 33587397

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited fom the Atlanta VA Medical Center in Atlanta, GA. Enrollment began in March 2013 and all study activities ended in March 15th, 2017. A total of 39 individuals were consented to participate in the study and passed screening, were randomly assigned to treatment arm and are included in the following results.
Pre-assignment Details: Two groups of participants were enrolled in the trial: Healthy controls and Schizophrenia subjects. The schizophrenia subjects were then randomized to either Oxytocin or Placebo.
  Note: for eye tracking and game outcomes, some subjects did not yield analyzable results due to the technical issues. Their data were therefore missing.
Groups:
- Healthy Controls: Participants having no psychiatric diagnosis were controls for this project. These controls will not receive oxytocin or placebo. They will only receive psychiatric screening interview, MATRICS Consensus Cognitive Battery (MCCB) assessment, urine drug screen, vision testing, and the three social cognition tasks.
- Oxytocin Arm: Participants receiving the intranasal oxytocin intervention received a dose of three 4 IU puffs per nostril for a total dose of 24 IU. Each puff is 0.1ml in volume so the total volume administered was 0.6 ml intranasally.
- Placebo Arm: Participants receiving the intranasal placebo intervention consisting of the OT vehicle administered as three puffs in each nostril. Each puff is 0.1ml in volume so the total volume administered will be 0.6 ml intranasally.
Period: Overall Study
Arm/Group | Healthy Controls | Oxytocin Arm | Placebo Arm
Started | 19 | 11 | 9
Completed | 19 | 11 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Oxytocin: Participants receiving the intranasal oxytocin intervention received a dose of three 4 IU puffs per nostril for a total dose of 24 IU. Each puff is 0.1ml in volume so the total volume administered was 0.6 ml intranasally.
- Placebo: Participants receiving the intranasal placebo intervention consisting of the OT vehicle administered as three puffs in each nostril. Each puff is 0.1ml in volume so the total volume administered will be 0.6 ml intranasally.
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Oxytocin | Placebo | Total
Number analyzed (Participants) | 19 | 11 | 9 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.36 (9.35) | 50.82 (9.16) | 47 (11.81) | 50.21 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 19 | 11 | 9 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 19 | 10 | 9 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 13 | 10 | 9 | 32
  White | 6 | 1 | 0 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 11 | 9 | 39
PANSS negative [Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Symptom Scale, negative symptom subscale. Contains 7 items, each with range of 1 to 7, to measure negative symptoms of schizophrenia. Total for this subscale ranges from 7 to 49. Higher score is worse.
  units on a scale | NA (NA) — The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. Healthy controls have no psychiatric diagnosis. | 13.64 (4.11) | 13.55 (4.25) | 13.6 (4.06)
PANSS positive [Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Symptom Scale, positive symptom subscale. Contains 7 items, each with range of 1 to 7, to measure positive symptoms of schizophrenia. Total for this subscale ranges from 7 to 49. Higher score is worse.
  units on a scale | NA (NA) — The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. Healthy controls have no psychiatric diagnosis. | 12.09 (2.62) | 11.55 (2.51) | 11.85 (2.52)
PANSS total [Mean (Standard Deviation); unit: units on a scale] — Positive and Negative Symptom Scale, total for whole scale. Contains 30 items, each with range of 1 to 7, to measure symptoms of schizophrenia. Total for this subscale ranges from 30 to 210. Higher score is worse.
  units on a scale | NA (NA) — The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. Healthy controls have no psychiatric diagnosis. | 49.18 (8.15) | 47.78 (7.41) | 48.55 (7.65)

OUTCOME MEASURES:

1. Primary Outcome: Eye Tracking: Fixation Count
Description: In order to assess the processing of social stimuli, subjects will be presented with a series of human faces of mixed sex and race showing neutral emotions and instructed to visually scan each face. Six regions of interest (ROIs) will be defined for each face stimulus: eyes, nose mouth, forehead, cheeks, and outside the contours of the face. The data will be processed off line for each face stimulus as the total time of fixation inside each of the ROIs. Refers to the number of fixations that occurred on the face of the stimulus presented to the participant during the eye-tracking assessment.
Time Frame: Day 1
Population: The analysis includes participants for which valid measurements are available: 16 participants in the Healthy Control Group, 11 in the Oxytocin Group and 9 in the Placebo Group.
Measure: Mean (Standard Deviation); unit: Number of face fixations
Arm/Group | Healthy Controls | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 11 | 9
Number of face fixations
  Eye Tracking-Gaze | 6.78 (3.74) | 9.19 (4.86) | 9.88 (4.83)
  Eye Tracking-Gender | 7.94 (4.90) | 8.34 (4.46) | 7.38 (6.24)

2. Primary Outcome: Eye Tracking: Dwell Duration Time
Description: Refers to the amount of time that an individual spent looking at the face of the stimulus presented to the participant during the eye-tracking assessment.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Healthy Controls | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 11 | 9
milliseconds
  Eye-Tracking Gaze | 1.11 (0.75) | 1.01 (0.57) | 1.18 (0.52)
  Eye-Tracking Gender | 1.26 (0.64) | 1.04 (0.66) | 0.99 (0.78)

3. Primary Outcome: Social Reward Ball-tossing Task
Description: Subjects will perform a computerized Social Reward Ball-Tossing Task in which they decide to return the ball to one of three fictional partners. The photos of the partners and their reciprocity in returning the ball to the subject will be manipulated. The number of balls sent to each of the partners will be quantified to assess socially reinforced learning. The result is expressed in number of ball tosses sent to the subject by a fictional player with a positive expression MINUS the number of ball tosses sent to the subject by a fictional player with a negative expression. These measures will be compared between the control subjects, oxytocin and placebo group.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of Ball tosses
Arm/Group | Healthy Controls | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 11 | 9
Number of Ball tosses | 8.91 (22.68) | 15.38 (29.19) | 25.64 (39.59)

4. Primary Outcome: Non-Social Reward Ball-tossing Game
Description: Social reward trials will be interleaved with non-social trials where subjects will play with random geometric shapes or landscape scenes associated with positive and negative non-social rewards. The outcome measure reported herein is the number of ball tosses the subject sends to shape A minus the number of ball tosses sent to shape B.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of ball tosses
Arm/Group | Healthy Controls | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 11 | 9
number of ball tosses | 10.53 (15.64) | 6.29 (15.69) | 28.20 (28.78)

5. Primary Outcome: Facial Emotion Identification Task
Description: The stimuli are 19 standard black and white pictures of faces showing one of six different emotions (happy, sad, angry, surprise, disgusted, ashamed) that were developed by Ekman and Friesen (1976). The pictures are shown for 15 sec, with 10 sec between each face. After the presentation of each face the subject is asked to choose which of the six emotions was displayed. The score on the test is the sum of correct responses. Subjects in the two groups (oxytocin vs. placebo) will be compared.
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Correct responses
Arm/Group | Healthy Controls | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 11 | 9
Correct responses | 12.16 (2.63) | 11 (3.58) | 9.44 (4.10)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the study Day 1 visit
Arm/Group | Healthy Controls | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 0/19 | 0/11 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-12-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT01568528/Prot_SAP_000.pdf